CLINICAL TRIAL: NCT04597957
Title: A Randomized Control Trial of a Fruit and Vegetable Prescription Program at a Federally Qualified Health System and Its Impact on Health Outcomes in Patients With Diabetes
Brief Title: The Fruit and Vegetable Prescription Program Study
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Collaborators: Blue Cross Blue Shield of Michigan Foundation (Other)
Responsible Party: Principal Investigator, Richard Bryce, Principal Invesigator, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10511
Record Dates: First submitted 2020-10-04; First posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fresh Rx Intervention group (Experimental): The Fresh Rx intervention group will receive up to 8 visits to the community based farmers market with $10 incentive for fruits and vegetables at each visit.
  Interventions: Dietary Supplement: Fresh Rx Intervention group
- Diabetic Standard of Care Control group (Active Comparator): Diabetic standard of care control group will receive no incentive for the community based farmers market.
  Interventions: Dietary Supplement: Fresh Rx Intervention group

INTERVENTIONS:
Dietary Supplement: Fresh Rx Intervention group — Fresh Rx Intervention participants will be able to fill their prescription at the FQHC based Farmers Market for fresh produce up to eight times during the 15-week Fresh Rx program. The provided debit cards will be loaded with the $10 stipend at each visit. At each market session, cooking demonstrations will take place that reinforce healthy food options and how to prepare foods that were available at the Mercado.
  All control group participants will be given flyers describing all the health and wellness programs at the FQHC including the Mercado. Control group participants will receive a $10 gift card to a national brand pharmacy (no fresh produce available). The enrollment time for the control group will overlap with the Fresh Rx group. After a 3-month time period, the control group will follow up and be given a $20 gift card to the same national brand pharmacy.

SUMMARY:
The Fruit and Vegetable Prescription Program Study is a pilot randomized controlled trial of patients with type 2 diabetes participating in a fruit and vegetable prescription program from a Federally Qualified Health Center in Detroit, MI . Changes in hemoglobin A1C (%), blood pressure (BP) and weight (lbs.) will be assessed changes to discern the impact on those that participated in a fruit and vegetable prescription program compared to those that received non-incentivized diabetes standard of care.

DETAILED DESCRIPTION:
Fresh Prescription (Fresh Rx) Program is a fruit and vegetable prescription program that brings together the healthcare system and the food system. This fosters innovative relationships to enhance the understanding of the correlation between food choices and health, increase consumption of locally grown fruits and vegetables, and build a healthy sustainable food system. This promising approach to a healthier food system connects patients to fresh, locally grown produce while providing direct economic benefits to small and midsize farmers and improving health and quality of life for participants.

The Fresh Rx program allots up to $80 ($10 per visit for up to eight visits) for purchase of fresh fruits and vegetables at that FQHC's farmers' market (referred to as the Mercado). The Mercado, which is located outside the entrance to the health center, is a collection of several local produce farmers. The Mercado operates every Thursday (9am-1pm) and will occur over 15 weeks from June 2018-October 2018. In addition to selling fresh produce, the Mercado also offers many other positive health promoting activities including cooking demonstrations, nutrition education and exercise events.

Fresh Rx participants are able fill their prescription at the Mercado for fresh produce up to eight times during the 15-week Fresh Rx program. The visits can, but do not necessarily need to be in consecutive weeks. The provided debit cards are loaded with the $10 stipend at each visit.

A list will be generated from the electronic medical records of the FQHC, of all non-pregnant patients with type 2 diabetes who had a HbA1C >8.0% over the 6 months prior to the start of the Fresh Rx Program. Using simple randomization, the list was randomized into two groups: The Intervention group and the control group. Those selected for the intervention group and the control group will be contacted by telephone and offered participation by a Community Health Worker. Once agreeable to participate, both groups will be brought into the center to sign an informed consent. At that time, they will have their BP, weight and HbA1C tested.

All Fresh Rx participants will complete a basic program orientation that includes receiving their Fresh Rx debit card that can be used with Mercado vendors. All participants will then have their BP, weight and HbA1C checked inside the FQHC after their last visit to the Mercado or within three months of the completion of the Fresh Rx program (January 2, 2019).

All control group participants will be given flyers describing all the health and wellness programs at the FQHC including the Mercado. No incentive will be given for the Mercado. Control group participants will be given a $10 gift card to a national brand pharmacy (no fresh produce available). The enrollment time for the control group will overlap the Fresh Rx group (June-September 2018). After a 3-month time period, control group participants will return and have a repeat BP, weight and HbA1C tested. They then will be given a $20 gift card to the same national brand pharmacy.

ELIGIBILITY:
Inclusion Criteria:

* FQHC patients with history of type 2 diabetics with a history of a hemoglobin a1c >8.0 % in the last 6 months.

Exclusion Criteria:

* individuals <18 years of age
* Pregnant patients
* type 1 diabetics
* those that decline participation in the Fresh Rx program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2018-07-12 (Actual); Primary Completion 2019-01-02 (Actual); Study Completion 2019-01-02 (Actual)

PRIMARY OUTCOMES:
Change in hemoglobin a1c (percent) of intervention and control group. | baseline, 3 months
  Both intervention and control groups will have hemoglobin a1c (%) tested at initial visit and 3 months after initial visit.
Change in systolic blood pressure (mmhg) of intervention and control group. | baseline, 3 months
  Both intervention and control groups will have systolic blood pressure (mmhg) tested at initial visit and 3 months after initial visit.
Change in diastolic blood pressure (mmhg) in intervention and control group. | baseline, 3 months
  Both intervention and control groups will have diastolic blood pressure (mmhg) tested at initial visit and 3 months after initial visit.
Change in weight (pounds) in intervention and control group. | baseline, 3 months
  Both intervention and control groups will have weight (pounds) tested at initial visit and and 3 months after initial visit.

SECONDARY OUTCOMES:
Number of visits to Clinic based farmers market (the mercardo) per participant in Fresh Rx program. | 15 weeks
  Fresh Rx participants were able fill their prescription at the Mercado for fresh produce up to eight times during the 15-week Fresh Rx program. The visits could, but did not necessarily need to be in consecutive weeks. The number of visits to the Mercado per participant will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Bryce, DO, Principal Investigator — Chass Center
Locations (2):
- United States (2):
  - Henry Ford Health System, Detroit, Michigan
  - Richard Bryce, Detroit, Michigan

IPD SHARING:
Plan to Share IPD: No